CLINICAL TRIAL: NCT02809079
Title: Mycophenolate Mofetil Treatment With Neuromyelitis Optica Spectrum Disorders in Chinese Patients
Acronym: MONICA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other); Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Wei Qiu, Associate Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016017
Record Dates: First submitted 2016-06-12; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Neuromyelitis Optica Spectrum Disorders; Mycophenolate Mofetil; Efficacy and Safety
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Mycophenolic Acid; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mycophenolate mofetil plus prednisone (Experimental): Mycophenolate mofetil 500mg Bid and prednisone 10mg Qd
  Interventions: Drug: Mycophenolate mofetil; Drug: Prednisone

INTERVENTIONS:
Drug: Mycophenolate mofetil — Mycophenolate mofetil 500mg Bid
Drug: Prednisone — prednisone 10mg Qd

SUMMARY:
Neuromyelitis optica (NMO) is an autoimmune inflammatory demyelinating disease of the central nervous system that leads to blindness and paralysis. Since disability accrues incrementally related to attacks, attack prevention with immunosuppressive therapy is the mainstay of preventing disability. However, there is no standard immunosuppressive treatment strategy for NMO relapse prevention. In a previous study, the investigators provided evidence supporting the use of azathioprine plus a low dose corticosteroid as an effective strategy which is associated with a reduction in the risk of relapse in Chinese patients with NMO, but azathioprine has bone marrow suppression and other side effects. Mycophenolate mofetil (MMF) is a new immunosuppressant with rapid onset, fewer side effects and other advantages. In recent years, MMF has been used in different immune-related neurological diseases; some literature shown the possible efficacy of MMF in NMO treatment.

In this research, a multi-center (Third Affiliated Hospital of Sun Yat-sen University, Zhongshan Ophthalmic Centre of Sun Yat-sen University, Nangfang Hospital of Southern Medical University) study will carry out to evaluate the efficacy and safety of mycophenolate mofetil therapy in NMO spectrum disorders.

ELIGIBILITY:
Inclusion Criteria:

* Meet the 2006 Wingerchuk diagnostic criteria;
* NMO-immunoglobulin G seropositive;
* Between 18 to 65 years old;
* Relapse: more than 2 relapses in recent 2 years; more than 1 relapses in recent 1 years;
* Expanded disability status scale: expanded disability status scale≤7.0, and visual acuity ≥20 / 100 at least in one eye
* Understand the purpose and procedures of this study, and written informed consent is obtained.

Exclusion Criteria:

* Using immunosuppressive agents and other drugs affect evaluation, and drug withdrawal less than 3 months;
* Patients with any of the following diseases: transaminases elevation exceed 2 times of the normal upper limit; white blood cell <4 × 109 / L, Hemoglobin <80g / L, platelet <100 × 109 / L;
* With serious cardiovascular, liver, kidneys and other vital organs and blood, endocrine system diseases, cancer history;
* With immunodeficiency, uncontrolled infection and active gastrointestinal diseases (such as gastric ulcer, etc.);
* Pregnancy, breast-feeding women and male or female who plans to conceive recently;
* Allergy to mycophenolate mofetil and prednisone.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Annualized relapse rate day 360 | day 360 after staring treatment
  Patients come back for follow-up visit on day 360 after staring treatment, and annualized relapse rate was evaluated.

SECONDARY OUTCOMES:
expanded disability status scale | day 1, 14, 30, 90, 180, 270, 360 after staring treatment
  Patients come back for follow-up visit on day 1, 14, 30, 90, 180, 270, 360 after staring treatment, and expanded disability status scale was evaluated.
Hauser scale | day 1, 14, 30, 90, 180, 270, 360 after staring treatment
  Patients come back for follow-up visit on day 1, 14, 30, 90, 180, 270, 360 after staring treatment, and Hauser scale was evaluated.
vision scale | day 1, 14, 30, 90, 180, 270, 360 after staring treatment
  Patients come back for follow-up visit on day 1, 14, 30, 90, 180, 270, 360 after staring treatment, and vision scale was evaluated.
Lesions in brain and spinal cord | day 1, 14, 30, 90, 180, 270, 360 after staring treatment
  Patients come back for follow-up visit on day 1, 14, 30, 90, 180, 270, 360 after staring treatment, lesions in brain and spinal cord were evaluated by MRI.
Annualized relapse rate | day 1, 14, 30, 90, 180, 270 after staring treatment
  Patients come back for follow-up visit on day 1, 14, 30, 90, 180, 270 after staring treatment, and annualized relapse rate was evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Qiu, Medical PhD, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: Yes
share by publications and meetings

REFERENCES:
- [Result] Falcini F, Trapani S, Ricci L, Resti M, Simonini G, de Martino M. Sustained improvement of a girl affected with Devic's disease over 2 years of mycophenolate mofetil treatment. Rheumatology (Oxford). 2006 Jul;45(7):913-5. doi: 10.1093/rheumatology/kei263. Epub 2006 Apr 25. No abstract available. PMID 16638802
- [Result] Huh SY, Kim SH, Hyun JW, Joung AR, Park MS, Kim BJ, Kim HJ. Mycophenolate mofetil in the treatment of neuromyelitis optica spectrum disorder. JAMA Neurol. 2014 Nov;71(11):1372-8. doi: 10.1001/jamaneurol.2014.2057. PMID 25199960
- [Result] Jacob A, Matiello M, Weinshenker BG, Wingerchuk DM, Lucchinetti C, Shuster E, Carter J, Keegan BM, Kantarci OH, Pittock SJ. Treatment of neuromyelitis optica with mycophenolate mofetil: retrospective analysis of 24 patients. Arch Neurol. 2009 Sep;66(9):1128-33. doi: 10.1001/archneurol.2009.175. PMID 19752302
- [Derived] Huang Q, Wang J, Zhou Y, Yang H, Wang Z, Yan Z, Long Y, Yin J, Feng H, Li C, Lu Z, Hu X, Qiu W. Low-Dose Mycophenolate Mofetil for Treatment of Neuromyelitis Optica Spectrum Disorders: A Prospective Multicenter Study in South China. Front Immunol. 2018 Sep 11;9:2066. doi: 10.3389/fimmu.2018.02066. eCollection 2018. PMID 30258442